CLINICAL TRIAL: NCT06673251
Title: Investigation of the Effects of Motor Performance, Sensory Processing, Quality of Life and Participation on School Readiness in Children with Type 1 Diabetes
Brief Title: School Readiness in Children with Type 1 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: arife akbulut (Other)
Responsible Party: Sponsor-Investigator, arife akbulut, LECTURER, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: AYBU-AKBULUT-002
Record Dates: First submitted 2024-08-14; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- children with type 1 diabetes
  Interventions: Other: motor and sensory assessments, surveys
- Healthy children
  Interventions: Other: motor and sensory assessments, surveys

INTERVENTIONS:
Other: motor and sensory assessments, surveys — It does not include any intervention. Only evaluation will be made.

SUMMARY:
It is known that motor and sensory functions are affected in children with type 1 diabetes (T1DM).This may cause children to have restrictions in their daily lives and decrease their participation in activities.Motor and sensory factors and participation are important factors affecting children's school readiness.This study was planned to investigate the effects of motor performance, sensory processing, quality of life and participation on school readiness in preschool children with T1DM.

ELIGIBILITY:
Inclusion Criteria:

Having been diagnosed with Type 1 DM in the last 6 months (for type 1 diabetes group) Being 60-78 months old

Exclusion Criteria:

* - Having any neurodevelopmental disorder in addition to diabetes (EX: cerebral palsy, down syndrome, muscular dystrophies..)
* Starting 1st grade

Ages: 60 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: TYPE 1 DİABETES CHİLDREN
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
school readiness | through study completion, an average of 1 year
  Marmara primary school school readiness scale (60-78 months)
  The scale consists of 2 forms:
  A. Development Form; It consists of a total of 153 behavioral items belonging to mental and language (74 items), socio-emotional (40 items), physical (23 items), self-care (16 items) skills.
  Each item is graded as "always, often, sometimes, never" to be filled by the teacher or parents according to the frequency of the child's behavior.
  B. Application Form; Mathematics (number recognition, increase-decrease, sets -color, shape-, ordering: 47 questions), Science (induction, deduction, problem solving: 14 questions), Sound (words starting with the same sound, rhyming words: 8 questions) Line (3 questions) Maze (2 questions) It consists of 5 sub-dimensions prepared to be answered by the child one-on-one in order to determine their success in their studies. Each question is scored (31) with (1) points for the correct answer and (0) points for the wrong answer.
motor performance | through study completion, an average of 1 year
  Bruininks-Oseretsky Motor Proficiency Test 2- (BOT 2) BOT 2 will be used to assess motor proficiency in children. BOT 2 is a test developed to assess fine and gross motor proficiency in children aged 4-21. The test duration can vary between 40 and 60 minutes for a child. The test consists of 8 subtests and 53 items. The maximum score that can be obtained from the test is 243. These are; fine motor skills (7 items - e.g.; Connecting the Dots), fine motor skill integrations (8 items - e.g.; Copying a Square), manual dexterity (5 items - e.g.; Classifying Shape Cards), bilateral coordination (7 items - e.g.; Sketch Jump), balance (9 items - e.g.; Walking on a Line), running speed and agility (5 items - e.g.; Sideways Jump on the Balance Beam), hand-arm coordination (7 items - e.g.; Dropping and Catching a Ball with Both Hands), strength (5 items - e.g.; Sit-up). A total motor composite score is also obtained from the total score of all items
Quality of Life | through study completion, an average of 1 year
  Pediatric Quality of Life Inventory (PedsQL)) PedsQL is a scale developed to measure the health-related quality of life of children and adolescents between the ages of 2-18. The PedsQL, which was developed for the ages of two to seven, was adapted into Turkish by Üneri and colleagues , and for the ages of 8-18 by Çakın, Memik and colleagues . PedsQL has only parent-report forms for children between the ages of 2-5, and both self-report and parent forms for children/adolescents between the ages of 5-18. PedsQL consists of 23 items.
Sensory Processing | through study completion, an average of 1 year
  The SPM Home Form consists of 75 items. The scale is evaluated with eight subscales: Social Participation, Vision, Hearing, Touch, Body Awareness, Balance and Movement, Planning and Ideas, and Total Sensory Systems in children aged 5-12. Total Sensory Systems represents the sum of the scores obtained from the Vision, Hearing, Touch, Body Awareness, Balance and Movement subscales and the Taste and Smell items, which are not subscales on their own. Each item is evaluated according to the frequency of the behavior with the expressions Never, Sometimes, Often, and Always. The Never option is given 1 point, the option is given 2 points, the option is given 3 points, and the option is given 4 points. Each item is related to a basic sensory integration sensitivity. In other words, the items can be interpreted as indicators of sensory overreactivity, underreactivity, sensory stimuli hunger, and a perception problem.
participation | through study completion, an average of 1 year
  The Participation and Environment Measure for Children and Youth (PEM-CY) questionnaire will be used. The PEM-CY is a parent-report questionnaire used to assess participation and environmental factors in home, school, and community settings among children and youth ages 5-17. The PEMCY participation items for each setting represent a broad range of activities typically performed in that setting. For each activity type, parents are asked (a) how often their child participates (never=0 to every day=7); (b) how involved their child is when participating (at least=1 to a lot=5); and (c) whether they would like a change in their child's participation (no or yes). Parents are then asked questions that include the PEM-CY environmental items for each setting. Information is collected about whether certain features of the environment help children participate in activities in that environment (no problem, usually helps, sometimes helps/sometimes makes it difficult, usually makes it difficult)

SECONDARY OUTCOMES:
physical fitness | through study completion, an average of 1 year
  The Munich Physical Fitness Test (MFUT) will be used to assess the physical fitness of children. The test consists of six different parameters including ball bouncing, target holding, forward bending, vertical jump, hanging and step test. After all parameters are completed, the score for each parameter is calculated from the standardization table appropriate for age and gender, and this total score is divided by six and recorded as the Munich score (20). MFUT has been shown to be a reliable and useful test in assessing important parameters of physical fitness such as strength, power, endurance, flexibility, speed, balance and coordination in children.

IPD SHARING:
Plan to Share IPD: No